CLINICAL TRIAL: NCT03613831
Title: Multi-center Complex Atrial Tachycardia High-Resolution Mapping Registry (MATH)
Status: Withdrawn | Type: Observational
Why Stopped: The sponsor has decided to stop the study
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PCR02
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Atrial Tachycardia (Including Atrial Flutter) Post Atrial Fibrillation Ablation or Cardiac Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: patient who used Rhythmia system and Orion catheter — suitable for Rhythmia system and Orion catheter according to relevant clinical guidelines and products instruction for use, per investigator's discretion

SUMMARY:
This study is an observational study without any hypothesis testing. It intended to observe the clinical application of electrophysiological mapping and catheter ablation of atrial tachycardia post atrial fibrillation ablation or cardiac surgery guided with Rhythmia System.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with atrial tachycardia (including atrial flutter) post atrial fibrillation ablation or cardiac surgery, which occurred at least 90 days prior to enrollment;
2. Subject is suitable for Rhythmia system and Orion catheter according to relevant clinical guidelines and products instruction for use, per investigator's discretion
3. Subject is age 18 or above;
4. Subject or his/ her legal representive understands and is willing to provide the Informed Consent Form (ICF) and participate in this trail.

Exclusion Criteria:

1. Subject with atrial fibrillation only;
2. Subject is enrolled in any other concurrent study that might interfere with this study;
3. Women of childbearing potential who are or might be pregnant at the time of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An arbitrary sample size of 100 should be enough for this registry study which may cover the focal, macro-reentry, micro-reentry and other types of atrial tachycardia. Assuming that the one-year recurrence rate post complex atrial tachycardia ablation is 30%, the 95% confidence interval of 100 samples shall be 21.2-40.0% (binomial distribution exact method).
  As per the current actual situation in China, it is predicted that 70-80 cases may be included for the atrial tachycardia post atrial fibrillation ablation, while 20-30 cases may be included for post cardiac surgery.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
target patient's type | 1 year
  Type of atrial tachycardia post atrial fibrillation ablation or cardiac surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China